CLINICAL TRIAL: NCT01814904
Title: A Multi-centre, Randomised, Controlled, Parallel Group, Open-label Study Evaluating the Efficacy, Safety and Tolerability of Three Doses of Colestilan (MCI-196) Compared to Standard Therapy With a Calcium-based Phosphate Binder, in Paediatric Subjects With Chronic Kidney Disease Stage 5 on Dialysis and With Hyperphosphataemia
Brief Title: Dose-finding Study of MCI-196
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study has been terminated because of insufficient patient recruitment.
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCI-196-E14
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Kidney Disease; Dialysis; Hyperphosphatemia; Paediatric
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MCI-196-L (Experimental): MCI-196 BSA eq 3g
  Interventions: Drug: colestilan-L
- MCI-196-M (Experimental): MCI-196 BSA eq 6g
  Interventions: Drug: colestilan-M
- MCI-196-H (Experimental): MCI-196 BSA eq 9g
  Interventions: Drug: colestilan-H
- CBPB (Active Comparator): Calcium-based P binder
  Interventions: Drug: CBPB

INTERVENTIONS:
Drug: colestilan-L — body surface area equivalent (BSAeq) 3 g/day
  Other Names: BindRen
  Arms: MCI-196-L
Drug: colestilan-M — BSAeq 6 g/day
  Other Names: BindRen
  Arms: MCI-196-M
Drug: colestilan-H — BSAeq 9 g/day
  Other Names: BindRen
  Arms: MCI-196-H
Drug: CBPB
  Arms: CBPB

SUMMARY:
The Primary Objective of this study is to determine the initial starting doses of colestilan (MCI-196) in paediatric subjects with Chronic Kidney Disease Stage 5 on Dialysis and with Hyperphosphataemia.

DETAILED DESCRIPTION:
This study has been terminated because of insufficient patient recruitment. There were no safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 years to <18 years with CKD stage 5 on dialysis (haemodialysis or peritoneal dialysis) for at least one month
* The subject has a documented diagnosis of hyperphosphataemia, as demonstrated by serum phosphorus(P) levels above the age-related upper limit of normal KDOQI Clinical Practice Guidelines for Nutrition in Children with CKD updated 2008)
* The subject has been taking CBPB prior to enrolment into the study (i.e., prior to the screening visit)
* The subject must have demonstrated serum P levels >1.5 standard deviation (SD) above the KDOQI 2008 age-related mean value at any time during the wash-out period (this must be demonstrated after stopping treatment with CBPB)
* At the time of randomisation, the subject must have demonstrated an increase in serum P levels from his/her most recent P central laboratory measurement by at least 10% above the pre-wash-out level

Exclusion Criteria:

* The subject has been diagnosed with hypocholesterolaemia (i.e., cholesterol levels below age-related normal ranges, per local practices)
* The subject has current clinically significant medical comorbidities, which may substantially compromise subject safety, or expose him/her to undue risk, or interfere significantly with study procedures and which, in the opinion of the Investigator, make the subject unsuitable for inclusion in the study (e.g., the subject currently has or has had a history of seizure disorders, dysphagia, swallowing disorders, predisposition to or current bowel obstruction, ileus or severe gastrointestinal [GI] disorders such as chronic or severe constipation [as judged by the Investigator], intestinal stenosis, intestinal diverticulum, sigmoid colitis, GI ulcers, current or a history of GI bleeding, or major GI tract surgery)
* The subject was treated with a combination of two or more phosphate binders within one month prior to screening
* The subject cannot stop treatment (prescription or over-the counter) of any of the following orally taken medications during the wash-out period: any product containing calcium (Ca), magnesium (Mg), aluminium compounds, sevelamer, lanthanum, ketosteril
* The subject is receiving immunosuppressant treatment for any medical condition at the time of randomisation or is expected to receive such treatment during the course of the study
* The subject is considered unstable on his/her current treatment for CKD within one month prior to screening (e.g., subjects starting treatment with vitamin D or its analogues, or other agents/procedures that may influence bone mineral metabolism [i.e., serum P and Ca levels])

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Mean absolute change in serum phosphorus | 17 weeks

SECONDARY OUTCOMES:
Proportion of responders (responders are defined as subjects demonstrating serum P levels ≤1.5 SD above the KDOQI 2008 age-related mean value) | 17 weeks
  Kidney Disease Outcomes Quality Initiative(KDOQI)
Mean absolute change in efficacy laboratory parameters (i.e.,P, Ca, Ca P ion product [CaxP], intact parathyroid hormone [iPTH], serum glucose, glycosylated haemoglobin [HbA1c], and uric acid) | 17 weeks
Mean percentage change in other efficacy laboratory parameters (i.e., lipid parameters [low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), total cholesterol, and triglycerides (TG)]) | 17 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site, London, United Kingdom